CLINICAL TRIAL: NCT00492128
Title: Comparative Trial of Combination Therapy of ARB/Diuretic Versus ARB/CCB in Uncontrolled Hypertensive Patients With Monotherapy of ARB
Brief Title: Kanagawa Combination Anti-hypertensive Therapy (K-CAT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Principal Investigator, Satoshi Umemura, Professor, Yokohama City University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200706001
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension
Keywords: hypertension; angiotensin receptor blocker; diuretic; combination therapy
MeSH Terms: conditions — Hypertension | interventions — Losartan; Amlodipine; hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan/hydrochlorothiazide (Experimental): Combination drug with losartan 50mg and hydrochlorothiazide 12.5mg
  Interventions: Drug: Losartan/amlodipine or losartan/hydrochlorothiazide
- Losartan/amlodipine (Active Comparator): Combination therapy with losartan 50mg and amlodopine 5mg
  Interventions: Drug: Losartan/amlodipine or losartan/hydrochlorothiazide

INTERVENTIONS:
Drug: Losartan/amlodipine or losartan/hydrochlorothiazide — Losartan 50mg/amlodipine 5mg and the fixed dose combination drug of losartan 50mg/hydrochlorothiazide 12.5mg once a day during 12 months.
  Other Names: Preminent (Hyzaar)

SUMMARY:
The purpose of this study is to compare the effect and safety of the antihypertensive combination therapies between losartan/amlodipine and fixed dose drug of losartan/hydrochlorothiazide.

DETAILED DESCRIPTION:
The combination therapy with multiple antihypertensive drugs is recommended in the patients who are uncontrolled with monotherapy. Diuretics increase the activities of renin-angiotensin-aldosterone system (RAS), and angiotensin receptor blockers (ARB) depress blood pressure potently in the state of increased RAS activities. Thus, the combination therapy with ARB and diuretics is expected to lower the blood pressure synergistically. This combination therapy is also expected to reduce the side effects of each drug. In this study, we will compare the effect and safety of the combination therapies between losartan/amlodipine and fixed dose drug of losartan/hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

* Under treatment of hypertension with ARB monotherapy for more than one month.
* systolic blood pressure more than 140mmHg and less than 160mmHg or diastolic blood pressure more than 90mmHg and less than 100mmHg in sitting position.
* In diabetic or CKD patients, systolic blood pressure more than 130mmHg and less than 160mmHg or diastolic blood pressure more than 80mmHg and less than 100mmHg in sitting position.

Exclusion Criteria:

* uncontrolled hypertension (diastolic blood pressure >120mmHg)
* uncontrolled diabetes mellitus (HbA1c>9.0%)
* Acute myocardial infarction, stroke and other cardiovascular events within six months
* The history of gout, or uric acid>8.0mg/dl
* Serum creatinine>2.0mg/dl
* sever liver dysfunction
* Bilateral renovascular stenosis
* secondary hypertension
* malignant hypertension
* uncontrolled arrhythmia
* pregnancy or possibility of pregnancy
* hypersensitivity to trial drug

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The change of systolic blood pressure | three months

SECONDARY OUTCOMES:
The achievement rate of target blood pressure | three months
The change of diastolic blood pressure | three months
The change of blood pressure | six months, nine months and one year
The achievement rate of target blood pressure | six months, nine months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Umemura, MD, PhD, Study Chair — Yokohama City University Graduate School of Medicine
Locations (1):
- Yokohama City University Graduate School of Medicine, Yokohama, Kanagawa, Japan